CLINICAL TRIAL: NCT03569969
Title: Comparison of Tympanoplasty Surgery Outcome Using Amniotic Membrane and Autologous Temporalis Fascia: A Randomized Clinical Trial Study
Brief Title: Comparison Tympanoplasty With Membrane Amniotic and Autologous Fascia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mohammad Sadegh Bagheri Baghdasht (Other)
Responsible Party: Sponsor-Investigator, Mohammad Sadegh Bagheri Baghdasht, Principal Investigator, Baqiyatallah Medical Sciences University
Organization: Baqiyatallah Medical Sciences University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ir.bmsu.rec.1395.233
Record Dates: First submitted 2018-01-11; First posted 2018-06-26 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Tympanic Membrane Perforation
Keywords: amniotic membrane; Tympanic Membrane Perforation
MeSH Terms: conditions — Tympanic Membrane Perforation | interventions — Tympanoplasty

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Experimental): Step1. Under local anesthesia and sedation , the temporal muscle fascia was removed, Step2. After the preparation on the tympanic membrane embedded , foam gel smeary with Dexamethasone was worn.Step3. Then the wound dressing was done with a gas number and a Surgifix. Step4. Patients were discharge from the operating room with an oral administration of Cephalexin capsules.
  Interventions: Procedure: Tympanoplasty With Autologous Fascia
- Test group (Experimental): Step1. After sedation and conducting local anesthesia with Lidocaine 2% and inserting the edges of the tympanic membrane and inserting the foam gel into the middle ear, amniotic membranes (produced in Iran tissue product) with a thickness of 100 microns on the tympanic membrane and the foam gel embedded. Step2. Under-layered and short-lived foam gel (manufactured by Ethicon Company) smeary with dexamethasone was covered.
  Interventions: Procedure: device: Tympanoplasty with Membrane Amniotic

INTERVENTIONS:
Procedure: device: Tympanoplasty with Membrane Amniotic — amniotic membrane Tympanoplasty
  Arms: Test group
Procedure: Tympanoplasty With Autologous Fascia — Autologous Temporalis fascia Tympanoplasty
  Arms: control group

SUMMARY:
The tympanic membrane separates the middle and the outer ear from each other and consists of three layers. The outer layer is covered with squamous epithelium, a thick basement membrane in the middle and an inner Mucosal layer. Rupture of the tympanic membrane is common cause of hearing loss.

In spite of the ability to spontaneously healing of the tympanic membrane, chronic tear of the eardrum in the absence of its spontaneously healing indicates surgical management. These surgeries are performing using various materials including fascia, cartilage, fats, pericardium and paper patch. It has proven that using different materials results in outcome and postoperative complications. The criteria of the best graft material includes availability, preservability, manageability, and acceptance rate to the hosts. Human amniotic membrane is preservable. Also, there isn't significant immunologic reactions against such graft material. So, choosing the best graft for Tympanoplasty surgery decreases complications, hospitalizations after surgery, and costs, consequently.

Up to now, limited studies have been conducted on the patients who were used amniotic membrane in the surgical reconstruction. There are different outcomes and complications which depend on the size of the rupture and the problems associated with the surgical conditions.

Considering that it can reduce the surgical time and cost of surgery, and with its high success rate, it can even be used as a substitute for conventional methods. The aim of this study was to compare the result of surgical repair of the tympanic membrane using membrane amniotic and surgical Tympanoplasty with Autologous fascia. Here the investigators reported on 30 patients who underwent Typmanoplasty with amniotic membrane and Temporalis fascia grafting.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Acute Otorrhea / - Cholesteatomas / - Canal stenosis requiring Canaloplasty / - Immunosuppressive patients / - Active neoplasm / - Diabetes Mellitus / - Ruptures less than one fifth of the eardrum / - Smoking.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Morbidity and surgical complications | Up to 1 year
  Signs and symptoms that are unexpectedly followed by surgery
The amount of restoration | Up to 1 year
  Restoration of tympanic membrane
Duration of hospitalization | 24 hour
  From the time of acceptance of the discharge

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Villar-Fernandez MA, Lopez-Escamez JA. Outlook for Tissue Engineering of the Tympanic Membrane. Audiol Res. 2015 Jan 23;5(1):117. doi: 10.4081/audiores.2015.117. eCollection 2015 Jan 21. PMID 26557361
- [Background] Catalano GB, Conticello S. [The long-term results of myringoplasty with amnion graft]. Otorinolaringologie. 1969 Apr-Jun;14(2):97-102. No abstract available. Romanian. PMID 5343906
- [Background] Harvinder S, Hassan S, Sidek DS, Hamzah M, Samsudin AR, Philip R. Underlay myringoplasty: comparison of human amniotic membrane to temporalis fascia graft. Med J Malaysia. 2005 Dec;60(5):585-9. PMID 16515109
- [Background] Rao TV, Chandrasekharam V. Use of dry human and bovine amnion as a biological dressing. Arch Surg. 1981 Jul;116(7):891-6. doi: 10.1001/archsurg.1981.01380190029007. PMID 7259490
- [Background] Silveira FC, Pinto FC, Caldas Neto Sda S, Leal Mde C, Cesario J, Aguiar JL. Treatment of tympanic membrane perforation using bacterial cellulose: a randomized controlled trial. Braz J Otorhinolaryngol. 2016 Mar-Apr;82(2):203-8. doi: 10.1016/j.bjorl.2015.03.015. Epub 2015 Sep 8. PMID 26631330
- [Background] Raj A, Sayal A, Rathore PK, Meher R. Sutureless tympanoplasty using acellular dermis. Am J Otolaryngol. 2011 Mar-Apr;32(2):96-9. doi: 10.1016/j.amjoto.2009.10.007. Epub 2010 Apr 13. PMID 20392523
- [Background] Hsu, G., Utilizing Dehydrated Human Amnion/Chorion Membrane Allograft in Transcanal Tympanoplasty. Otolaryngology, 2014. 4(161): p. 2.
- [Background] Ghanavati SZ, Shousha MA, Betancurt C, Perez VL. Combined conjunctival autograft and overlay amniotic membrane transplantation; a novel surgical treatment for pterygium. J Ophthalmic Vis Res. 2014 Jul-Sep;9(3):399-403. doi: 10.4103/2008-322X.143386. PMID 25667744